CLINICAL TRIAL: NCT06965452
Title: Trans Arterial Embolization for Facet Arthropathy
Brief Title: Trans-arterial Embolization for the Treatment of Facet Pain Due to Facet Arthropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-1020
Record Dates: First submitted 2025-04-23; First posted 2025-05-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Facet Joint Arthropathy; Pain; Osteoarthritis
Keywords: Facetogenic pain; Facet pain; Facet joint pain; Low back pain; Back Pain
MeSH Terms: conditions — Pain; Osteoarthritis; Low Back Pain; Back Pain | interventions — Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: The intervention consists of a trans-arterial injection of the vascular supply the facet joints using Embozene microspheres. After patients have failed conservative management with proven facetogenic pain they will be enrolled into the study. Patients will be brought to the neurointerventional suite and have a diagnostic spinal angiogram under procedural sedation. The dorsal segmental arteries supplying the facet joints causing back pain will be embolized using Embozene microspheres approved particles.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Embozene Microspheres for Facetogenic Low Back Pain (Experimental): This is a single site, single arm study to assess the safety and efficacy of trans arterial embolization using Embozene microspheres of the facet joint for the treatment of facetogenic low back pain.
  Interventions: Device: Spinal angiography and embolization/ Embozene Microspheres

INTERVENTIONS:
Device: Spinal angiography and embolization/ Embozene Microspheres — Once consent is obtained the patient will be scheduled for spinal angiography and embolization. The patient will undergo the procedure at North Shore University Hospital. After embolization the patient will be monitored in recovery for 5 hours and then discharged to home.
  The primary objective of this study is to examine the safety and feasibility of trans arterial embolization of the facet joint using Embozene Microspheres for the treatment of back pain from facet arthropathy and osteoarthritis.

SUMMARY:
This single-site, single-arm study evaluates the feasibility, safety, tolerability, and efficacy of trans-arterial embolization (TAE) using Embozene microparticles for treating facetogenic pain due to facet arthropathy (osteoarthritis of the facet joints) in the lumbar spine.

DETAILED DESCRIPTION:
This is a single site, single-arm study assessing the feasibility, safety, tolerability, and efficacy of trans-arterial embolization for the treatment of facet pain due to facet arthropathy. Osteoarthritis is a common and major cause of pain and disability. Each spinal level contains multiple joints including the intervertebral discs as well as the facet joints. Degeneration of the facet joints or facet arthritis begins early in life and the prevalence grows with increasing age ultimately reaching as high as 100% in people over 60 years of age. Facet arthritis can lead to the development of facetogenic pain. Previous studies have suggested that trans-arterial embolization may be beneficial for pain in the setting of osteoarthritis. Trans-arterial injections have been described in the knee, hip, and shoulder.

Embolization of the dorsal branches of the segmental arteries supplying the bony elements of the spine is a well-established technique employed for preoperative embolization of bony spinal tumors and metastatic disease. Previous studies have clearly demonstrated safety of the techniques with low overall risk. In one large series of 100 embolizations there was only one recorded complication due to the embolization. However, it has not been described for use in the setting of facet arthropathy (OA of the facet joint). The PI for this study has published the results of large series of embolization for spinal tumors without any serious adverse events. Currently the treatment of lumbar spine OA involved medical management, followed by minimally invasive techniques such as intraarticular injection and neurolysis, which are of questionable efficacy, and ultimately possible spinal surgery and fusion in the setting of degenerative disease and structural abnormalities. The purpose of this study is to demonstrate the safety and preliminary efficacy of trans-arterial facet joint embolization using Embozene microparticles in patients with facet arthropathy and lumbar spine OA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85

  * Confirmed diagnosis of spinal facet arthropathy on MRI OR CT
  * Confirmed diagnosis of lumbosacral facetogenic pain based on diagnostic nerve blocks.
  * Failed medical management of pain.

    * Back pain persistent for at least 6 months
    * Pain worse than at least 6/10 on a visual analog pain scale
  * Failed at least one of either intra-articular injections of steroids/ anesthetics or neuro-ablative procedure.
  * Maximum of 2 spinal levels of facetogenic pain in the lumbar and sacral spine (i.e. L4-5 and L5-S1).
  * Modified Rankin Scale 0-2

Exclusion Criteria:

* - Pregnancy
* History of prior spinal embolization at the target level.
* History of surgery/ stenting of the aorta at the level of embolization.
* Severe allergic reaction to iodinated contrast (i.e. anaphylaxis)
* Creatinine > 1.5 mg/dl and/or creatinine clearance < 60 mL/min (except if patients is already on hemodialysis).
* Modified Rankin Scale >2
* Angiographic/ Procedural Exclusion Criterion: Vascular supply to the spinal cord from the vessels supplying the facet joints targeted for embolization.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Procedure-Related Serious Adverse Events in the Perioperative Period | 1 year
  The primary outcome measurements for safety are:
  -The number of procedure-related serious adverse events occurring in the perioperative period

SECONDARY OUTCOMES:
Proportion of Patients with >20% Improvement in Facetogenic Pain Based on Visual Analog Scale (VAS). Percent from 0% to 100% and higher % represents greater improvement. | 1 year
  Secondary endpoints include:
  - >20% improvement of facetogenic pain based on visual analog pain scale before and after the procedure
Proportion of Patients with >20% Improvement in Disability Based on Oswestry Low Back Pain Disability Questionnaire | 1 year
  Secondary endpoints include:- >20% improvement in disability based on Oswestry Low Back Pain Disability Questionnaire.Percent from 0% to 100% and higher % represents greater improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States